CLINICAL TRIAL: NCT01029938
Title: Comparative Study of Covered Stent With Coil Embolization in the Treatment of Cranial Internal Carotid Artery Aneurysm: A Nonrandomized Prospective Trial
Brief Title: Treatment of Cranial Internal Carotid Artery Aneurysm With Willis Covered Stent and Coil Embolization
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Cerebral aneurysm study in China, The Sixth Affiliated People's Hospital, Shanghai Jiao Tong University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASC2; SAPH002
Record Dates: First submitted 2009-12-08; First posted 2009-12-10 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2009-12

CONDITIONS: Intracranial Aneurysms
Keywords: Intracranial aneurysms;; Covered stent;; Coil embolization
MeSH Terms: conditions — Intracranial Aneurysm | interventions — p80-coilin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Covered stent (Active Comparator): The Willis covered stent specifically designed for intracranial vasculature was developed by our institution and the MicroPort Medical Company (Shanghai, China), and coil embolization, which has been widely applied for nearly two decades, is currently the endovascular approach that is first recommended for intracranial aneurysm treatment.
  Interventions: Procedure: Covered stent; Procedure: Coil
- Coil (Active Comparator): Coil embolization, which has been widely applied for nearly two decades, is currently the endovascular approach that is first recommended for intracranial aneurysm treatment.
  Interventions: Procedure: Covered stent; Procedure: Coil

INTERVENTIONS:
Procedure: Covered stent — Consecutive patients with CICA aneurysms were endovasculartreated with a Willis covered stent (group A) or coil embolization (group B)
  Other Names: GDCs, covered stent
Procedure: Coil — Consecutive patients with CICA aneurysms were endovasculartreated with a Willis covered stent (group A) or coil embolization (group B)
  Other Names: GDCS, covered stent

SUMMARY:
Intracranial aneurysm treatment with coil embolization is associated with relatively low complete occlusion and high recanalization rates. The investigators evaluate whether Willis covered stent implantation yields angiographic and clinical results superior to those with coil embolization.

DETAILED DESCRIPTION:
Endovascular treatment of intracranial aneurysms with detachable coils has been widely used since the introduction of GDCs in 1991 and has been proven to be effective in preventing rebleeding after aneurysmal rupture. The clinical and angiographic results of endovascular coil occlusion of intracranial aneurysms are positive, with an initial and final overall complete occlusion rate of 35.9%-76.8% and 38.3%- 87.8%. In the mid- and long-term, however, aneurysm recanalization may occur in as many as one-third of cases.

The natural history of aneurysm recurrence after coil treatment is often benign, but bleeding from incompletely coiled aneurysms is a well-documented threat, moreover, the degree of aneurysm occlusion after treatment was strongly associated with risk of rerupture. Even if 100% occlusion of the aneurysms after the initial treatment was obtained on immediate postembolization angiography, there was still a relatively high recanalization rate (26.4%) on long-term follow-up angiography. In a recent study, we have confirmed that there was still aneurysm perfusion of the aneurysm sac in a complete occluded aneurysm no matter on initial or follow-up rotate digital angiography. In addition, some authors have demonstrated that endothelialization of the aneurysm orifice following placement of GDCs can occur; however, it appears to be the exception rather than the rule.

To overcome these disadvantages, the Willis covered stent, specially designed for intracranial vasculature, has been developed by our institution and the MicroPort Medical Company (Micro-Port, Shanghai, China). Our preliminary results demonstrated good flexibility and efficacy of the Willis covered stent in the treatment of cranial internal carotid artery aneurysms (CICA) in patients without an extremely tortuous ICA (Radiology 2009; 253:470-7), and also the covered stents have been proved to be more effective than re-coiling with regard to complete occlusion of recurrent aneurysms (J Neurol Neurosurg Psychiatry 2009;16:[Epub ahead of print]). Since 2005, we have performed a nonrandomized prospective trial of endovascular treatment CICA aneurysms with a covered stenting or coil embolization. So, we evaluate whether implantation of a primary Willis covered stent yielded angiographic and clinical results that superior to those with the currently recommended approach of coil embolization.

ELIGIBILITY:
Inclusion Criteria:

1. Definite CICA aneurysm, either ruptured or unruptured, as demonstrated by arterial angiography;
2. Parent artery diameter of 3.0-5.0 mm;
3. Good tolerance of BOT; and
4. At least one control angiogram taken > 6 months after the initial treatment

Exclusion Criteria:

1. An extremely tortuous vessel proximal to the parent artery and/or lack of appropriate accessible routes, thereby rendering the patient unsuitable for endovascular treatment;
2. Parent artery diameter of < 3 mm or > 5.0 mm;
3. Inability of the patient to undergo general anesthesia or endovascular intervention; or
4. Expected patient survival of < 1 year because of other co-existing diseases. -

Ages: 10 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2005-04; Primary Completion 2008-09 (Actual); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Willis covered stent indicate good flexibility and efficacy in cranial internal carotid artery (CICA) aneurysm treatment in patients without an extremely tortuous ICA | 53 months after the study

SECONDARY OUTCOMES:
Willis covered stents are more effective than recoiling with respect to the complete occlusion of recurrent aneurysms | 56 months after the study

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated People's Hospital, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Li MH, Li YD, Tan HQ, Luo QY, Cheng YS. Treatment of distal internal carotid artery aneurysm with the willis covered stent: a prospective pilot study. Radiology. 2009 Nov;253(2):470-7. doi: 10.1148/radiol.2532090037. Epub 2009 Sep 29. PMID 19789235
- [Result] Li YD, Li MH, Gao BL, Fang C, Cheng YS, Wang W, Li WB, Zhao JG, Zhang PL, Wang J, Li M. Endovascular treatment of recurrent intracranial aneurysms with re-coiling or covered stents. J Neurol Neurosurg Psychiatry. 2010 Jan;81(1):74-9. doi: 10.1136/jnnp.2009.171967. Epub 2009 Aug 16. PMID 19687026
- [Derived] Li MH, Leng B, Li YD, Tan HQ, Wang W, Song DL, Tian YL. Comparative study of covered stent with coil embolization in the treatment of cranial internal carotid artery aneurysm: a nonrandomized prospective trial. Eur Radiol. 2010 Nov;20(11):2732-9. doi: 10.1007/s00330-010-1854-z. Epub 2010 Aug 11. PMID 20700595